CLINICAL TRIAL: NCT03693456
Title: An Exploratory Pilot Study Evaluating the Correlation Between Conjunctival Allergen Challenge (CAC) Response to Dissolved Food Allergen and Previously Performed Oral Escalating Dose Food Challenge Response
Brief Title: Food Allergy Diagnostic Test Response to Previous Oral Challenge Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: ORA-FA-002
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2016-02

CONDITIONS: Food Hypersensitivity
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Responders Without Epinephrine (Experimental): Subjects experienced a positive response during previous oral food challenge without a severe adverse event and did not require epinephrine. Will be subjected to a conjunctival allergen challenge.
  Interventions: Other: Conjunctival Allergen Challenge
- Responders With Epinephrine (Experimental): Subjects experienced a positive response during previous oral food challenge and required epinephrine. Will be subjected to a conjunctival allergen challenge.
  Interventions: Other: Conjunctival Allergen Challenge
- Non-Responders (Experimental): Subjects did not experience a positive response during previous oral food challenge. Will be subjected to a conjunctival allergen challenge.
  Interventions: Other: Conjunctival Allergen Challenge

INTERVENTIONS:
Other: Conjunctival Allergen Challenge — Food allergen dissolved in water will be instilled in an increasing titrated fashion into the subjects eye and response will be graded according to proprietary scales.

SUMMARY:
The objective of this study is to compare the ocular response to CAC (using food allergen sensitive patients) to the systemic response of a previously performed oral food allergen challenge in the same subjects. This study will investigate the potential utility of CAC as a predictive tool for identifying patient response to food allergen challenge and maximum tolerated dose.

DETAILED DESCRIPTION:
Patients usually discover they have food allergies after consuming a given food and experiencing a subsequent allergic reaction. The majority of patients (75%) will then consult a food allergist for formal diagnosis and treatment information.1 With respect to patient quality of life, there is tremendous benefit in having a confirmed diagnosis of food allergy as often patients are unsure of the source of their reaction outside the office. Allergists will conduct Skin Prick Test (SPT) and assess serum specific IgE levels to screen for specific food protein sensitivities. However, a positive response in SPT and specific IgE will confirm only sensitivity, and in more than 70% of cases patients that respond positively to SPT and specific IgE testing will NOT manifest an allergic response to food consumption.2 To address this issue, most food allergists will recommend an oral food challenge in a controlled setting to confirm the allergic response from consuming the suspected foods. The oral food challenge (OFC) consists of consuming escalating levels of the suspect food, (usually mixed in applesauce or controlled baked goods), until either a reaction manifests or until the challenge is complete with no reaction. The food challenge process poses significant risk to the patient. In 5% of cases, the patient experiences a severe allergic response which requires the use of epinephrine.2,3 These responses typically consist of severe reactions in GI or respiratory and arise from challenging patients with higher doses of food allergen then is necessary to prove a mild allergic response. The reason an allergist would give an increased dose that the patient reacts to with severity results from misdiagnosing the mild forms of the reaction during the titrated challenge. It is this shortcoming in diagnosis that could be addressed by identifying high-risk patient populations through conjunctival allergen challenge and through the development of additional objective diagnostic endpoints.

We hypothesize that conjunctival allergen challenge (CAC) may be able to predict which patients are likely to experience an adverse event during a food allergen challenge. The appearance of severe ocular response following CAC (level II on a 0-2 Scale) has been shown to correlate well with a positive food response during escalating food challenge, and represented a better predictor of food allergen than skin test and serum specific IgE combined.4 We hypothesize that the severity of the ocular response to CAC titration, or the appearance of related non-ocular signs and symptoms of systemic response to CAC (itchy palate, wheezing, FEV1 reduction) could correlate with the likelihood of experiencing a severe adverse event during food challenge. In order to mitigate the occurrence of severe adverse events during food challenge, and to determine if the CAC response can serve as a useful tool for informing the clinician of anticipated patient response patterns to oral food allergen challenge, we will perform CAC titration on a population of food allergy patients that previously underwent oral food escalating challenge. Any patterns in CAC response will be compared to historical food allergen reactivity and occurrence of severe adverse responses to evaluate the potential of the CAC as a predictive tool that could add value to the oral food challenge model.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female of any race, at least 5 years of age with documented food challenge in the past 12 months;
* Have provided verbal and written informed consent. If under 18, a parent/guardian must provide consent for the subject;
* Negative pregnancy test for women of childbearing potential;
* Be willing and able to follow instructions, including participation in study assessments, and can be present for the required study visits for the duration of the study;

Exclusion Criteria:

* Be a woman who is pregnant or nursing an infant;
* Be unable to discontinue short-acting antihistamines for three days or long-acting antihistamines for five to seven days (depending on half-life) prior to CAC;
* Have asthma that has evolved and now fulfills any of the criteria defined as follows:

  1. uncontrolled persistent asthma by National Asthma Education and Prevention Program Asthma guidelines (2007) or by Global Initiative for Asthma (2011) or being treated with combination therapy of medium dose inhaled corticosteroid with a long acting inhaled β2-agonists.
  2. at least two systemic corticosteroid courses for asthma in the past year or one oral corticosteroid course for asthma in the past three months.
  3. prior intubation for asthma in the past year;
* Be receiving β-blocking agents, angiotensin-converting enzyme inhibitors, angiotensin-receptor blockers, calcium channel blockers or tricyclic antidepressant therapy;
* Be receiving or planning to receive anti-tumor necrosis factor drugs or anti-IgE drugs (such as omalizumab) or any biologic immunomodulatory therapy;
* Be receiving or planning to receive any type of immunotherapy to any food (e.g. oral immunotherapy, sublingual immunotherapy, specific oral tolerance induction) during their participation in the study;
* Be receiving or planning to receive any aeroallergen immunotherapy during their participation in the study;
* Be suffering from generalized dermatologic disease (e.g. severe atopic dermatitis, uncontrolled generalized eczema, ichthyosis vulgaris);
* Have any new disorder in which epinephrine is contraindicated such as coronary artery disease, uncontrolled hypertension, or serious ventricular arrhythmias;
* Have experienced severe anaphylaxis resulting in emergency hospitalization;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Ora Calibra Ocular Itching Scale | Ten minutes after each CAC dose through duration of challenge (up to 90 minutes)
Ora Calibra Ocular Hyperemia Scale | Ten minutes after each CAC dose through duration of challenge (up to 90 minutes)
Ora Calibra Itchy Palate/Mouth Scale | Ten minutes after each CAC dose through duration of challenge (up to 90 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Maeve E O'Connor, M.D., Principal Investigator — Allergy, Asthma & Immunology Relief (AAIR) of Charlotte
Locations (1):
- Allergy, Asthma & Immunology Relief (AAIR) of Charlotte, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No